CLINICAL TRIAL: NCT00012142
Title: Randomized, Double-Blind, Placebo-Controlled, Phase II Study Of Intravenous CCI-779 Administered Weekly To Patients With Androgen-Independent Prostate Cancer
Brief Title: CCI-779 in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068487; UCLA-000606401; GENE-C9940-32; UCLA-CCI-779; W-AR-3066K1-201-US; NCI-G01-1917
Record Dates: First submitted 2001-03-03; First posted 2004-03-26 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2002-05

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — temsirolimus

INTERVENTIONS:
Drug: temsirolimus

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to determine the effectiveness of CCI-779 in treating patients who have progressive prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of CCI-779 in patients with androgen-independent prostate cancer. II. Determine the effects of CCI-779 on prostate-specific antigen levels in these patients. III. Assess the pharmacokinetic parameters of CCI-779 in these patients. IV. Assess the possible pharmacodynamic relationship of CCI-779 with clinical response in these patients. V. Determine the impact of CCI-779 on the quality of life in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 4 arms. Arm I: Patients receive low-dose CCI-779 IV over 30 minutes weekly. Arm II: Patients receive high-dose CCI-779 IV over 30 minutes weekly. Arm III: Patients receive low-dose placebo IV over 30 minutes weekly. Arm IV: Patients receive high-dose placebo IV over 30 minutes weekly. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who develop progressive disease while receiving placebo may cross over to the equivalent dose of CCI-779. Quality of life is assessed at baseline; at weeks 4, 8, 12, 24, and 36; and at final/cross-over visit. Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed asymptomatic, progressive, metastatic adenocarcinoma of the prostate Progressive disease defined as increasing prostate-specific antigen (PSA) levels from 2 measurements at least 2 weeks apart PSA greater than 5 ng/mL Continued medical means of gonadal ablation (e.g., luteinizing hormone releasing hormone (LHRH)) required No known CNS metastases unless previously treated by surgery or radiotherapy and stable, asymptomatic, and not requiring steroids and anticonvulsants

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 6 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8.5 g/Dl Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST no greater than 3 times ULN (no greater than 5 times ULN if liver metastases present) Serum cholesterol no greater than 350 mg/Dl Triglycerides no greater than 300 mg/Dl Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No unstable angina or life-threatening ventricular arrhythmia requiring maintenance therapy No myocardial infarction within the past 6 months Other: No other malignancy in past 5 years other than basal cell or squamous cell skin cancer HIV negative No active infection Not immunocompromised No other major illness that would preclude study Fertile patients must use effective contraception during and for 3 months after the study

PRIOR CONCURRENT THERAPY: Biologic therapy: Concurrent epoetin alfa allowed Chemotherapy: No prior cytotoxic chemotherapy for prostate cancer No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 6 weeks since prior antiandrogen therapy At least 4 weeks since prior hormonal therapy (6 weeks for antiandrogens) for prostate cancer other than continued LHRH agonist No concurrent systemic corticosteroids No concurrent anticancer hormonal therapy Radiotherapy: At least 3 weeks since prior radiotherapy No prior palliative radiotherapy to more than one site No prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium No concurrent radiotherapy Surgery: At least 3 weeks since prior surgery Other: At least 4 weeks since prior investigational agent No concurrent immunosuppressive agents No other concurrent investigational agent No concurrent enzyme-inducing anticonvulsants (carbamazepine, phenobarbital, phenytoin), ketoconazole, diltiazem, rifampin, terfenadine, cisapride, astemizole, or pimozide No concurrent megestrol acetate for appetite Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Prager, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States